CLINICAL TRIAL: NCT03089203
Title: Phase I Study of CART-PSMA-TGFβRDN Cells in Patients With Advanced Castrate Resistant Prostate Cancer
Brief Title: CART-PSMA-TGFβRDN Cells for Castrate-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 32816, 826250
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): CART-PSMA-TGFβRDN cells 1-3x10^7 Day 0
  Interventions: Biological: CART-PSMA-TGFβRDN cells
- Cohort 2 (Experimental): CART-PSMA-TGFβRDN cells 1-3x10^8 Day 0
  Interventions: Biological: CART-PSMA-TGFβRDN cells
- Cohort -3 (Experimental): CART-PSMA-TGFβRDN cells 1-3x10^7 Day 0
  Interventions: Biological: CART-PSMA-TGFβRDN cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort 4 (Experimental): CART-PSMA-TGFβRDN cells 0.70-1.00 x 10^8 Day 0
  Interventions: Biological: CART-PSMA-TGFβRDN cells; Drug: Cyclophosphamide; Drug: Fludarabine
- Cohort 3 (Experimental): CART-PSMA-TGFβRDN cells at the MTD (established by Cohorts 1-2) on day 0
  Interventions: Biological: CART-PSMA-TGFβRDN cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CART-PSMA-TGFβRDN cells — autologous CAR T cells
Drug: Cyclophosphamide — 300 mg/m2/day given over 3 days
  Arms: Cohort -3; Cohort 3; Cohort 4
Drug: Fludarabine — 30 mg/m2/day given over 3 days
  Arms: Cohort -3; Cohort 3; Cohort 4

SUMMARY:
This is a single center, single arm Phase I study to establish the safety and feasibility of intravenously administered lentivirally transduced dual PSMA-specific/ TGFβ-resistant CAR modified autologous T cells (CART-PSMA-TGFβRDN cells) in patients with metastatic castrate resistant prostate cancer.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety and feasibility of lentivirally transduced PSMA-TGFβRDN autologous CAR T cells administered with and without cyclophosphamide/fludarabine lymphodepleting chemotherapy in a 3+3 dose escalation design. Subjects must receive the dose of CART-PSMA-TGFβRDN cells as per their cohort assignment in order to be considered evaluable for DLT assessments at that dose level. Subjects who do not receive CART-PSMA-TGFβRDN cells as per their cohort assignment will not be evaluable for DLT assessments/MTD determination, however they will still be followed per protocol and will be included in the overall safety analysis, as well as the analysis of secondary and exploratory endpoints. Subjects who enroll but do not receive CART-PSMA-TGFβRDN cells will be removed from the study and replaced.

Up to 5 dosing cohorts will be explored as follows:

* Cohort 1 subjects (N=3 or 6): will receive a single dose of 1-3 x 107/m2 lentivirally transduced CART-PSMA-TGFβRDN cells on day 0 without any conditioning chemotherapeutic regimen. If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level. If 0 DLT/3 subjects or 1 DLT/6 subjects occurs, the study will advance to Cohort 2. If 2 DLT/3 subjects occurs at dose of 1-3 x 107/m2 cells, then enrollment in this Cohort will be stopped and the dose will be de-escalated by 10-fold to 1-3 x 106 cells/m2 (Cohort -1). In this situation, up to 6 subjects will be enrolled in Cohort -1.
* Cohort 2 subjects (N=3 or 6): will receive a single dose of 1-3 x 108/m2 lentivirally transduced CART-PSMA-TGFβRDN cells on day 0 without any conditioning chemotherapeutic regimen. If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level. If 0 DLT/3 subjects or 1 DLT/6 subjects occurs, the study will advance toIf 2 DLT/3 subjects occur, then the study will stop and declare maximum tolerated dose (MTD).

Cohorts 1 and 2 were originally designed to identify the MTD of CART-PSMA-TGFβRDN cells. The highest dose level where only 0/3 or 1/6 DLTs were observed in a given cohort will be defined as the MTD for evaluation in Cohort 3.

COHORT 3 CLOSED WITH PROTOCOL V10

* Cohort 3 subjects (N=3 to 9): will receive a single dose of lentivirally transduced CART-PSMA-TGFβRDN cells at the MTD (established by Cohorts 1-2) on day 0, following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given over 3 days; lymphodepleting chemotherapy will be scheduled such that the last day of chemotherapy is 3 days (± 1 day) prior to the infusion of CART-PSMA-TGFβRDN cells. This treatment regimen will be evaluated as follows:

  * If 0 DLT /3 subjects occur, the study will enroll an additional 6 patients to confirm further evaluate the safety of this treatment regimen.
  * If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level to further evaluate safety. If 1 DLT/6 subjects and the safety of this treatment regimen is established, another 3 subjects may be enrolled to further evaluate the safety of this treatment regimen.
  * If 2 DLT/3 subjects or 2 DLT/6 subjects occurs, then enrollment into this cohort will be stopped and the CART-PSMA-TGFβRDN dose will be de-escalated to 1x107/m2 CART-PSMA-TGFβRDN cells with lymphodepleting chemotherapy (Cohort -3). At least 3 subjects would be treated in the Cohort -3 de-escalation cohort.
* Cohort -3 subjects (N=3 to 6): will open in the event of unacceptable toxicity in Cohort 3. Subjects enrolled into this cohort will receive a single dose of 1-3 x 107/m2 lentivirally transduced CART-PSMA-TGFβRDN cells on day 0, following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given over 3 days; lymphodepleting chemotherapy will be scheduled such that the last day of chemotherapy is 3 days (± 1 day) prior to the infusion of CART-PSMA-TGFβRDN cells. Up to 6 subjects will be treated in this dose de-escalated cohort to demonstrate the safety of this regimen.

Once the safety of the Cohort -3 dosing regimen has been established, a new dose escalation Cohort 4 will be opened to enrollment. The 1st three infusions in Cohort 4 will be staggered by 28 days to allow for the assessment of DLTs. If no safety concerns are identified in the first three subjects within this cohort, subsequent infusions within Cohort 4 will be staggered by at least 14 days.

• Cohort 4 subjects (N=3 to 6): Subjects enrolled into this cohort will receive a single dose of 0.70-1.00 x 108 lentivirally transduced CART-PSMA-TGFβRDN cells on Day 0, following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given over 3 days. Lymphodepleting chemotherapy will be scheduled such that the last day of chemotherapy is 3 days (± 1 day) prior to the infusion of CART-PSMA-TGFβRDN cells.

* If 1 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level. If 1 DLT/6 subjects occurs, this dose level will be established as safe; and the safety of the CART-PSMA-TGFβRDN cells may continue to be further explored as part of a subsequent expansion amendment.
* If 0 DLT/3 subjects occurs, the study will enroll an additional 3 subjects at this dose level to further evaluate safety. If 0 DLT/6 subjects or 1 DLT/6 subjects occurs, this dose level will be established as safe; and the safety of the CART-PSMA-TGFβRDN cells may continue to be further explored as part of a subsequent expansion amendment. .
* If 2 DLTs occur at any time, enrollment in this cohort will be stopped and the study will be paused for additional investigation.

At the investigator's discretion, subjects may receive "retreatment" with CART-PSMA-TGFβRDN cells at any point after Day 28, provided that safety of the cohort-defined treatment regimen has been established.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic castrate resistant prostate cancer
2. ≥10% tumor cells expressing PSMA as demonstrated by immunohistochemistry analysis on biopsied tissue. RETIRED WITH PROTOCOL VERSION 15
3. Radiographic evidence of osseous metastatic disease and/or measurable, non-osseous metastatic disease (nodal or visceral)
4. Patients ≥ 18 years of age
5. ECOG performance status of 0 - 1
6. Adequate organ function, as defined by:

   1. Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 cc/min
   2. Serum total bilirubin < 1.5x ULN
   3. Serum ALT/AST < 2x ULN
7. Adequate hematologic reserve within 4 weeks of eligibility confirmation by physician-investigator as defined by:

   1. Hgb > 10 g/dl
   2. PLT > 100 k/ul
   3. ANC > 1.5 k/ul Note: Subjects must not be transfusion dependent
8. Evidence of progressive castrate resistant prostate adenocarcinoma, as defined by:

   1. Castrate levels of testosterone (< 50 ng/ml) with or without the use of androgen-deprivation therapy AND
   2. Evidence of one of the following measures of progressive disease in the 12 weeks preceding eligibility confirmation by physician:

   i. soft tissue progression by RECIST 1.1 criteria ii. osseous disease progression with 2 or more new lesions on bone scan (as per PCWG2 criteria) iii. increase in serum PSA of at least 25% and an absolute increase of 2 ng/ml or more from nadir (as per PCWG2 criteria)
9. Prior therapy with at least one standard initial therapy for the treatment of metastatic castrate resistant prostate cancer (i.e. docetaxel chemotherapy, 17α lyase inhibitor, or second-generation anti-androgen therapy)
10. Provides written informed consent
11. Subjects of reproductive potential must agree to use acceptable birth control methods

Exclusion Criteria:

1. Treatment with immune checkpoint inhibitors and immunoconjugate therapies, including nivolumab, pembrolizumab, atezolizumab, ipilimumab, and/or durvalumab, within 2 months prior to eligibility confirmation by physician-investigator. Cancer vaccine therapies (such as Sipuleucel-T or PROSTVAC) are allowable as a prior line of therapy. Radium-223 is allowable as a prior line of therapy, provided laboratory complete blood counts meet all inclusion criteria as above, without transfusion support in the preceding 4 weeks.
2. History of an active non-curative non-prostate primary malignancy within the prior 3 years
3. Subjects with a rising PSA, but who have never had radiologic evidence of metastatic disease (i.e. 'biochemical recurrence') RETIRED WITH PROTOCOL VERSION 6
4. Subjects who require the chronic use of systemic corticosteroid therapy. Patients may be on a low dose of steroids (≤10mg equivalent of prednisone).
5. Subjects who have received > 4 prior therapies for the treatment of castrate resistant prostate cancer (excluding luteinizing hormone-releasing hormone agonists or antagonists, or first generation anti-androgen therapies). Note: Docetaxel or abiraterone/prednisone administered in the castration-sensitive setting will count as a prior line of therapy. RETIRED WITH PROTOCOL V13
6. Subjects with Class III/IV cardiovascular disability according to the New York Heart Association Classification
7. Subjects with symptomatic vertebral metastases affecting spinal cord function (as determined by clinical history, physical exam, or MRI imaging)
8. Active autoimmune disease, including connective tissue disease, uveitis, inflammatory bowel disease, or multiple sclerosis; or a history of severe (as judged by the physician-investigator) autoimmune disease requiring prolonged immunosuppressive therapy
9. Patients with ongoing or active infection.
10. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
11. Active hepatitis B, hepatitis C or HIV infection.
12. Active medical condition that, in the opinion of the physician-investigator, would substantially increase the risk of uncontrollable CRS or CAR Neurotoxicity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2038-09-08 (Estimated); Study Completion 2038-12-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events, laboratory toxicities and clinical events that are possibly, likely, or definitely related to study participation. | 15 years
  using CTCAE v 4.03
Clinical feasibility is defined as the frequency of subjects enrolled on this protocol who do not receive CART-PSMA-TGFβRDN cells. | 30 days
Manufacturing feasibility is determined by the frequency of product release failures and the occurrence of dose failures (inability to meet target dose). | 30 days

SECONDARY OUTCOMES:
Assess the clinical anti-tumor effect of CART-PSMA-TGFβRDN cells by RECIST | 6 months
  RECIST 1.1 criteria for soft tissue disease
Assess the clinical anti-tumor effect of CART-PSMA-TGFβRDN cells by PCWG2 | 6 months
  PCWG2 criteria for osseous disease
Assess the clinical anti-tumor effect of CART-PSMA-TGFβRDN cells by serum PSA measurement | 6 months
  serum PSA measurement
Assess the clinical anti-tumor effect of CART-PSMA-TGFβRDN cells by overal survival (OS). | 15 Years
Assess the clinical anti-tumor effect of CART-PSMA-TGFβRDN cells by number of subjects with progression free survival (PFS). | 15 Years

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Haas, MD, Principal Investigator — Universtiy of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Narayan V, Barber-Rotenberg JS, Jung IY, Lacey SF, Rech AJ, Davis MM, Hwang WT, Lal P, Carpenter EL, Maude SL, Plesa G, Vapiwala N, Chew A, Moniak M, Sebro RA, Farwell MD, Marshall A, Gilmore J, Lledo L, Dengel K, Church SE, Hether TD, Xu J, Gohil M, Buckingham TH, Yee SS, Gonzalez VE, Kulikovskaya I, Chen F, Tian L, Tien K, Gladney W, Nobles CL, Raymond HE; Prostate Cancer Cellular Therapy Program Investigators; Hexner EO, Siegel DL, Bushman FD, June CH, Fraietta JA, Haas NB. PSMA-targeting TGFbeta-insensitive armored CAR T cells in metastatic castration-resistant prostate cancer: a phase 1 trial. Nat Med. 2022 Apr;28(4):724-734. doi: 10.1038/s41591-022-01726-1. Epub 2022 Mar 21. PMID 35314843
- [Derived] Kloss CC, Lee J, Zhang A, Chen F, Melenhorst JJ, Lacey SF, Maus MV, Fraietta JA, Zhao Y, June CH. Dominant-Negative TGF-beta Receptor Enhances PSMA-Targeted Human CAR T Cell Proliferation And Augments Prostate Cancer Eradication. Mol Ther. 2018 Jul 5;26(7):1855-1866. doi: 10.1016/j.ymthe.2018.05.003. Epub 2018 May 8. PMID 29807781